CLINICAL TRIAL: NCT04606940
Title: Study of Circulating Tumor DNA (ctDNA) Kinetics in Immuno-oncology: Intense Dynamic Monitoring of ctDNA in Advanced/Metastatic Head and Neck Squamous Cell Carcinoma (HNSCC) Patients Treated With Immune Checkpoint Inhibitors.
Brief Title: Study of Circulating Tumor DNA (ctDNA) Kinetics in Immuno-oncology (IO-KIN)
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Other Study IDs: IO-KIN; 20-5803 (Other: CAPCR ID)
Record Dates: First submitted 2020-10-18; First posted 2020-10-28 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Head and Neck Cancer; Advanced Cancer; Metastatic Cancer; HNSCC; Squamous Cell Carcinoma
Keywords: Head and Neck; Immune Checkpoint Inhibitors; Immuno-oncology; Liquid Biopsy; Advanced Cancer; Metestatic Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasm Metastasis; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Squamous Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples collected serially for cfDNA and gDNA extraction. Archived tumor sample collected for tumor genomic DNA analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IO-KIN: Patients with a histological or cytological confirmed recurrent, metastatic or advanced HNSCC of the oral cavity, oropharynx, hypopharynx, larynx or unknown origin (but being treated as HNSCC). Patients who are going to receive at least one dose of anti-PD1 antibody (nivolumab or pembrolizumab).

SUMMARY:
This study aims to study the kinetics of ctDNA levels after the first dose of immune checkpoint inhibitor in patients with recurrent or metastatic head and neck cancer. This is an important study to understand the optimal timing for ctDNA quantitation for future studies in immunotherapy, though further validation would be needed in other tumor types. It may help standardize the most relevant blood collection time points so that patients will not be subjected to multiple blood draws at random time points in future liquid biopsy trials.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytological confirmed recurrent, metastatic or advanced HNSCC of the oral cavity, oropharynx, hypopharynx, larynx or unknown origin (but being treated as HNSCC).
* Availability of tumor sample.
* Patients who are going to receive at least one dose of anti-PD1antibody (nivolumab or pembrolizumab).

Exclusion Criteria:

* Nasopharynx, maxillary sinus, nasal/nasal vestibule squamous tumors
* Patients who are receiving concomitantly any other tumor-specific treatment (chemotherapy, radiotherapy, any monoclonal antibodies different from anti- PD-1 antibodies).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of advanced/metastatic head and neck squamous cell carcinoma (HNSCC) of the oral cavity, oropharynx, hypopharynx or larynx or unknown origin (but being treated as HNSCC) and are receiving at least one dose of nivolumab or pembrolizumab.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2021-10-12 (Actual); Study Completion 2021-10-12 (Actual)

PRIMARY OUTCOMES:
The change in kinetics of ctDNA changes in advanced/metastatic will be measured for HNSCC patients treated with immune checkpoint inhibitors (anti-PD-1 antibody). | Through study completion, up to 1.5 years
  At each time-point, absolute ctDNA levels will be calculated from all test targets (including undetected targets).The change in ctDNA from baseline to every time-point is defined as the percentage change in absolute ctDNA levels in plasma at that end point since baseline.

SECONDARY OUTCOMES:
The changes in ctDNA levels will be measured. These value will help correlate with progression free survival (PFS) and overall survival (OS). | Through study completion, up to 1.5 years
  At each time-point, absolute ctDNA levels will be calculated from all test targets (including undetected targets).The change in ctDNA from baseline to every time-point is defined as the percentage change in absolute ctDNA levels in plasma at that end point since baseline.
The optimal time-point will be measured to analyze ctDNA as a predictive marker of response to immune checkpoint inhibitors (anti-PD-1 antibody). | Through study completion, up to 1.5 years
  At each time-point, absolute ctDNA levels will be calculated from all test targets (including undetected targets).The change in ctDNA from baseline to every time-point is defined as the percentage change in absolute ctDNA levels in plasma at that end point since baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Siu, Principal Investigator — Princess Margaret Cancer Centre; Scott Bratman, Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Targeted gene sequencing results, along with limited clinical information that does not identify the patient as an individual, such as age, partial date of birth (year, month), gender, cancer type, and pathology information related to the samples tested, and survival time may be shared with collaborating researchers.
  Data from this study can be shared through two types of databases: open-access or controlled-access. An open-access database is publicly accessible and contains limited clinical information and analyses of samples. A controlled-access database contains more detailed clinical information, such as relevant past medical history and the results of prior and ongoing cancer treatments, and analyses of samples, but is only accessible to researchers who sign agreements defining how data may be used. All data will be stripped of all personal identifying information.